CLINICAL TRIAL: NCT05161637
Title: A Phase 2/3, Randomized, Double-blind, Comparator- and Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Efficacy of TLC590 for Postsurgical Pain Management Following Inguinal Hernia Repair
Brief Title: Phase 2/3 Study of TLC590 for Postsurgical Pain Management
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLC590A2003
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Postsurgical Pain Management
MeSH Terms: interventions — Bupivacaine; Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TLC590 490mg (Experimental): TLC590 490mg (20mL)
  Interventions: Drug: TLC590
- TLC590 588mg (Experimental): TLC590 588mg (24mL)
  Interventions: Drug: TLC590
- Bupivacaine 75mg (Active Comparator): Bupivacaine HCl 75mg (30mL)
  Interventions: Drug: Bupivacain
- Ropivacaine (Active Comparator): Ropivacaine HCl 150mg (30mL) (Part 1)
  Interventions: Drug: Ropivacaine
- Normal saline (Placebo Comparator): Normal Saline 0.9% (20mL or 24mL)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: TLC590 — TLC590 490mg or 588mg
  Other Names: intestigational drug
  Arms: TLC590 490mg; TLC590 588mg
Drug: Bupivacain — Bupivacaine 75mg
  Other Names: active comparator
  Arms: Bupivacaine 75mg
Drug: Ropivacaine — Ropivacaine 150mg
  Other Names: active comparator
  Arms: Ropivacaine
Drug: Normal saline — Normal saline 20mL or 24mL
  Other Names: placebo
  Arms: Normal saline

SUMMARY:
A phase 2/3 randomized, double-blind, 2-part, comparator- and placebo-controlled study to assess the safety, pharmacokinetics and efficacy of postsurgical local infiltration in adult subjects following inguinal hernia repair surgery.

DETAILED DESCRIPTION:
This is a phase 2/3 randomized, double-blind, 2-part, comparator- and placebo-controlled study to assess the safety, pharmacokinetics and efficacy of postsurgical local infiltration in adult subjects following inguinal hernia repair surgery. This study includes 2 parts. An unblinded interim analysis will be performed after completion of part 1 (phase 2, approximately 115 subjects to be randomized for 2 different doses of TLC590, bupivacaine, ropivacaine, or placebo), for selecting a TLC590 dose for part 2 (phase 3, approximately 300 subjects to be randomized for TLC590, bupivacaine, or placebo).In this study, 2 doses of TLC590 24.5 mg/mL in inguinal hernia repair will be assessed in an initial phase 2 part before proceeding to a phase 3 pivotal evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* BMI 18-39 kg/m2
* Scheduled to undergo a primary, unilateral Lichtenstein inguinal hernia repair with mesh
* ASA Physical Status Classification of 1, 2 or 3

Exclusion Criteria:

* Clinically significant abnormal clinical laboratory test value
* Clinically significant 12-lead ECG
* History of orthostatic hypotension or syncope
* History of significant renal, hepatic, gastrointestinal, cardiovascular, metabolic, neurologic, psychiatric, or other condition
* History of seizure or currently taking anticonvulsants
* History of hypersensitivity to bupivacaine/ropivacaine, any other amide-type local anesthetic, propofol, oxycodone or morphine (or other opioids)
* History of severe or refractory post-operative nausea or vomiting (PONV)
* Abnormalities of laboratory parameters: HbA1c, platelet, hemoglobin, WBC, serun bilirubin/alanine aminotransferase/aspartate aminotrasferase, serum creatinine, PTT/INR
* Concurrent acute, or chronic painful restrictive/physical condition
* Received opioid therapy for longer than 4 days per week
* Prohibited medication: aspirin and other anti-platelet medication, anticoagulants, class III antiarrhythmic drugs, strong CYP1A2 inhibitors,systemic corticosteroids, NSAID, opioid, bupivacaine or ropivacaine, any investigational product
* History of drug abuse or alcohol abuse
* Positive results on the urine drug screen or alcohol breath test
* History of HIV; active HBV or HCV
* An inguinal hernia repair in the last 3 months or has undergone 3 or more surgeries within 12 months
* Malignancy in the last 2 years
* Documented sleep apnea or on home continuous positive airway pressure treatment (CPAP)
* Personal or family history of malignant hyperthermia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Part 1 - AUC 0-24 of NPRS-M | 0-24 hours
  AUC 0-24 of NPRS-M, evaluated comparing each dose of TLC590 with Placebo
Part 2 - AUC 0-72 of NPRS-M | 0-72 hours
  AUC 0-72 of NPRS-M, evaluated comparing each dose of TLC590 with Placebo

SECONDARY OUTCOMES:
AUC 0-72 of NPRS-M (active comparator) | 0-72 hours
  AUC 0-72 of NPRS-M (TLC590 vs Bupivacaine)
Proportion of opioid-free subjects through 72 hours (placebo) | 0-72 hours
  Proportion of opioid-free subjects through 72 hours (TLC590 vs. Placebo)
Proportion of opioid-free subjects through 72 hours (active comparator) | 0-72 hours
  Proportion of opioid-free subjects through 72 hours (TLC590 vs. Bupivacaine)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Tai, PhD, Study Director — Taiwan Liposome Company

IPD SHARING:
Plan to Share IPD: No